CLINICAL TRIAL: NCT03953807
Title: A 12-month, Prospective, Open-label, Phase 4 Study to Evaluate the Efficacy and Safety of OZURDEX® (Dexamethasone Intravitreal Implant) in Treatment Naïve Patients (According to Standard Clinical Practice) With Diabetic Macular Edema
Brief Title: A Study to Evaluate the Effectiveness and Safety of OZURDEX® in Patients With Diabetic Macular Edema But Never Treated
Acronym: EYEberia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-MA-EYE-0603; 2018-004785-33 (EudraCT Number)
Record Dates: First submitted 2019-05-13; First posted 2019-05-17 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ozurdex (Experimental): OZURDEX implant 700 μg
  Interventions: Drug: Dexamethasone Intravitreal Implant

INTERVENTIONS:
Drug: Dexamethasone Intravitreal Implant — Implant 700 μg

SUMMARY:
This study will evaluate the efficacy and safety of OZURDEX in patients with Diabetic Macular Edema when used in a real world setting in Spain and Portugal.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of diabetes mellitus (type 1 or type 2)
* Media clarity, pupillary dilation, and patient cooperation sufficient for all study procedures
* Written informed consent obtained in accordance with all local privacy requirements

Exclusion Criteria:

* Uncontrolled systemic disease
* History of disease, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease condition that contraindicates the use of the investigational drug, might affect the interpretation of study results, or render the patient at high risk from treatment complications
* Patients who have been previously treated for DME (two focal laser allowed)
* Untreated diabetes or anticipated change (increase) of antidiabetic medications during the study
* Elevated IOP or glaucoma diagnosis
* Any active ocular infection or inflammation
* Aphakia
* A substantial cataract is present that is likely to be decreasing visual acuity by three lines or more (i.e., cataract would be reducing visual acuity to 20/40 or worse if the eye was otherwise normal)
* Anticipated need for ocular surgery during the study
* History of vitrectomy or incisional glaucoma surgery - Female patients who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using a reliable means of contraception
* Known allergy, hypersensitivity or contraindication to the study medication, its components, or povidone iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Mean change in best corrected visual acuity (BCVA) 2 months (± 2 weeks) after the last injection | Baseline, at Month 10 through 12

SECONDARY OUTCOMES:
Mean change in Central Retinal Thickness (CRT) 2 months (± 2 weeks) after the last injection received | Baseline, at Month 10 through 12
Mean retreatment interval in months | During the 12 to 14-month study
Area under the curve (AUC) for CRT | Baseline, During the 12 to 14-month study
AUC for BCVA | Baseline, During the 12 to 14-month study
Mean change in the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25) | Baseline, at Month 14
  25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Original numeric values from the survey will be recoded with the worst and best possible scores set at 0 and 100 points, respectively. In this format, scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score.
Proportion of patients with 2nd injection | During the 12 to 14-month study
Proportion of patients with 3rd injection | During the 12 to 14-month study
Mean number of injections administered | During the 12- to 14-month study
Time to 3rd injection | During the 12 to 14-month study
Time to 2nd injection | During the 12 to 14-month study

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (26):
- Portugal (6):
  - Chuc /Id# 233643, Coimbra
  - Hospital de Santo Andre /ID# 233670, Leiria
  - IRL - Instituto de Retina e Diabetes Ocular de Lisboa /ID# 233667, Lisbon
  - Centro Hospitalar de Lisboa Norte /ID# 233684, Lisbon
  - Ulsam /Id# 233635, Viana do Castelo
  - Hospital de Vila Franca de Xira /ID# 233682, Vila Franca de Xira
- Spain (20):
  - Instituto Oftalmológico Gómez-Ulla /ID# 233590, Santiago de Compostela, A Coruna
  - Hospital Universitari Son Espases /ID# 233601, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Puerta de Hierro, Majadahonda /ID# 233597, Majadahonda, Madrid
  - CLINICA UNIVERSIDAD DE NAVARRA-Pamplona /ID# 233618, Pamplona, Navarre
  - Centro de Oftalmología Barraquer /ID# 233591, Barcelona
  - ICOF Hospital Clinic De Barcelona /ID# 233675, Barcelona
  - Instituto de Microcirugía Ocular /ID# 233689, Barcelona
  - Hospital Universitario de Cruces /ID# 233673, Bilbao
  - Hospital Universitario Insular de Gran Canaria /ID# 233658, Les Palma
  - Oftalvist Moncloa /ID# 233647, Madrid
  - Vissum Madrid /ID# 233646, Madrid
  - Hospital Clinico Universitario San Carlos /ID# 233578, Madrid
  - Hospital Universitario La Paz /ID# 233619, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 233609, Seville
  - Hospital General Universitario de Valencia /ID# 233600, Valencia
  - Hospital Universitario Arnau Vilanova /ID# 233594, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 233613, Valencia
  - Hospital Universitario de Araba /ID# 233693, Vitoria-Gasteiz
  - Hospital Clinico Universitario Lozano Blesa /ID# 233685, Zaragoza
  - Miguel Servet University Hospital /ID# 233629, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance.,To be considered as a site for current and futur — http://www.AllerganClinicalTrials.com